CLINICAL TRIAL: NCT06130449
Title: The Role of Androgens in Neurophysiological and Autonomic Function in Male Veterans With Spinal Cord Injury
Brief Title: Testosterone and Neural Function
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: B5028-M; 1IK1RX005028-01 (NIH)
Record Dates: First submitted 2023-10-25; First posted 2023-11-14 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; testosterone; cardiovascular; neurophysiology; central nervous system; autonomic; motor function; electrical stimulation; cardiovagal function
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Participant-blinded crossover placebo-controlled pilot study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participant-blinded (Ayr Saline Gel)
  Interventions: Drug: Ayr Saline Nasal Gel
- Intranasal TRT (Active Comparator): Participant-blinded (11 mg of Natesto)
  Interventions: Drug: Natesto testosterone intranasal gel

INTERVENTIONS:
Drug: Natesto testosterone intranasal gel — A single dose of Natesto (11 mg total, 5.5 mg per nostril) will be administered to each participant.
  Other Names: testosterone intranasal gel
  Arms: Intranasal TRT
Drug: Ayr Saline Nasal Gel — A single dose of Ayr (one spray per nostril) will be administered to each participant.
  Other Names: Saline Nasal Gel
  Arms: Placebo

SUMMARY:
Spinal cord injury (SCI) disrupts the nerves controlling movement, along with those that regulate functions like heart rate and blood pressure (known as the autonomic nervous system, or ANS). Testosterone (T) plays a significant role in brain health and ANS reflex function in non-neurologically impaired men. However, little is known about the relationships between T, nerve function, and ANS dysfunction after SCI. Interestingly, up to 60% of men with SCI exhibit persistently low T concentrations, which may worsen nerve and ANS dysfunction. In uninjured eugonadal people (normal physiologic range of serum T concentrations), a single pharmacologic dose of intranasal T has been shown to quickly improve nerve function, but no study has evaluated if T administration alters nerve and ANS function in men with SCI. Herein, the investigators will conduct the first study to test how a single dose of intranasal T impacts motor and ANS function in this population.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) disrupts sensorimotor function and corticospinal excitability, resulting in muscle weakness and autonomic nervous system (ANS) dysfunction that detracts from cardiovascular (CV) health. These deficits may be exacerbated by low testosterone (T), which develops in most men during the acute/subacute phases of SCI and persists in 45-60% of men thereafter. Low T (hypogonadism) is associated with multiple health impairments, including reduced lean tissue mass and increased fat mass, systemic inflammation, and risk for CV and neurodegenerative diseases. Moreover, low T is associated with CV ANS dysfunction and impaired cardiovagal (parasympathetic) reflex function following SCI. In men with low T after SCI, restoring T concentrations to the normal (eugonadal) range with T replacement therapy (TRT) improves energy expenditure, body composition, CV function, and markers of cardiometabolic health. Evidence from animal models also demonstrates that T is neuroprotective, upregulates neurotrophic factors, and promotes neuroplasticity and myelin regeneration. However, the neural effects of intranasal TRT are unknown.

T is the most abundant bioactive androgen within the circulation. It exerts direct biological actions by binding androgen receptors (ARs), affecting transcription, as well as non-genomic mechanisms in the brain, spinal cord, heart, and numerous other tissues throughout the body. The majority of circulating T is bound to sex-hormone binding globulin (SHBG) and albumin, with only 1-4% circulating unbound (free T). Free T and albumin-bound T are collectively termed bioavailable T, as SHBG-bound T cannot readily dissociate to engage cellular receptors. In this regard, a high prevalence of men with SCI not only exhibit low total T, but also exhibit a marked reduction in bioavailable T because there is a >10-fold increase in SHBG after SCI, resulting in lower proportions of free and albumin-bound T.

The primary goal of this proposal is to perform a small pilot/feasibility study to assess neurophysiological and cardiovagal responses to a single dose of intranasal TRT in a cohort of these men who exhibit low Total T (<300 ng/dL), low Free T (<46 pg/mL), or low bioavailable T (<110 ng/dL) and hypogonadal signs/symptoms.

Primary Aim: To investigate the acute effects of a single dose of intranasal TRT (11 mg) compared with placebo on CNS excitability and cardiovagal reflex function 30 minutes after administration in 15 male Veterans (10 with chronic SCI and 5 uninjured controls) who have low baseline total T concentrations. CNS excitability will be assessed using hand muscle electromyography (EMG) output determined by recruitment curves evoked by non-invasive single-pulse transcranial magnetic stimulation (TMS) and cervical transcutaneous spinal cord stimulation (TSCS). A cold face challenge (CFC) while measuring beat-to-beat heart rate signals will be used to examine CV ANS reflex function. Because this Exploratory Aim is a pilot/feasibility study, formal hypothesis testing would be premature. However, based on the literature, the investigators expect that elevating circulating concentrations of T into the high normal physiologic range via intranasal TRT will result in improved neural and cardiovagal function for 6-8 hours after the dose.

The results of this pilot study will inform feasibility and identify modifications needed to design a larger eventual trial to evaluate the efficacy and safety of intranasal TRT. Ours will be the first clinical study to collect pilot/feasibility data on an intranasal TRT formulation that has the potential to improve neural function after SCI. This is significant because our results are expected to provide evidence demonstrating the feasibility of a novel intranasal therapeutic strategy in Veterans with SCI.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Hypogonadal (Serum Total T <300 ng/dL, Free T <46 pg/mL, or bioavailable T <110 ng/dL) with signs/symptoms of hypogonadism
* Age 18-80 years
* Traumatic or non-traumatic spinal cord injury (SCI)
* Time since injury (TSI) more than 12 months
* American Spinal Injury Association (ASIA) Injury classification Scale (AIS) A, B, C, or D
* Stable prescription medication regimen for at least 30 days
* Not currently receiving pharmacological treatment for hypogonadism
* Must be able to commit to study requirements of 3 visits within a 30-day period
* Provide informed consent

Exclusion Criteria:

* Extensive history of seizures
* Ventilator dependence or patent tracheostomy site
* History of neurologic disorder other than SCI
* History of moderate or severe head trauma
* Currently receiving treatment for hypogonadism
* History of allergy, hypersensitivity, or other significant adverse reaction to testosterone replacement therapy
* Significant cardiovascular disease or cardiac conduction disease
* Active psychological disorder
* Moderate or severe brain injury, stroke, tumor, multiple sclerosis, or abscess
* Recent history (within 3 months) of substance abuse
* Pressures sores stage 3 or greater
* Active infection
* Frequent severe migraines
* Recent history (within past 6 months) of recurrent autonomic dysreflexia, defined as a syndrome of sudden rise in systolic pressure greater than 20 mm Hg or diastolic pressure greater than 10 mm Hg, without rise in heart rate, accompanied by symptoms such as headache, facial flushing, sweating, nasal congestion, and blurry vision (this will be closely monitored during all screening and testing procedures)
* History of implanted devices with electromagnetic properties: brain/spine/nerve stimulators, aneurysm clips, ferromagnetic metallic implants in the head (except for inside mouth); cochlear implants; cardiac pacemaker/defibrillator; intracardiac lines; currently increased intracranial pressure; or other contraindications to brain or spine stimulation
* Use of medications that significantly lower seizure threshold, such as amphetamines, neuroleptics, dalfampridine, and bupropion.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Electromyographic (EMG) responses | up to one day
  Response to electrical and magnetic stimulation, singly, will be measured via peak-to-peak amplitude (millivolts) in first dorsal interosseous and abductor pollicis brevis muscles.

SECONDARY OUTCOMES:
Serum Testosterone | up to one day
  Serum testosterone will be assessed prior to and after administration of intranasal TRT.
Cardiovagal Function (heart rate variability) | up to one day
  Changes in beat-by-beat heart rate (beats per minute) signals collected using ECG during a cold face challenge (cardiovagal provocation) to determine cardiovagal reflex function. Changes in the high frequency (0.15-0.4 Hz) component will be used as an indication of parasympathetic activity to the heart.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob A Goldsmith, PhD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No